CLINICAL TRIAL: NCT01825083
Title: The Effect of Ketamine in the Prevention of Hypoventilation in Patients Undergoing Deep Sedation Using Propofol and Fentanyl
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in personnel
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Gildasio De Oliveira, Prinipal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STU00068533
Record Dates: First submitted 2013-01-31; First posted 2013-04-05 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Hypercarbia
Keywords: Hypercarbia; TOSCA monitor; Ketamine; Fentanyl; Intraoperative monitoring
MeSH Terms: conditions — Hypercapnia | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine (Active Comparator): Ketamine administered 0.5mg/kg followed by an infusion of 1.5mcg/kg/min.
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): Saline group will received the same volume in saline as the ketamine dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — Ketamine group receives 0.5mg/kg followed by an infusion of 1.5mcg/kg/min.
  Other Names: Ketamine adminstration
  Arms: Ketamine
Drug: Placebo — 0.9 % normal saline group receives same volume as the ketamine dose
  Other Names: 0.9 % normal saline group receives same volume as ketamine dose
  Arms: Placebo

SUMMARY:
Procedures performed under sedation have the same severity in regards to morbidity and mortality as procedures performed under general anesthesia1. The demand for anesthesia care outside the operating room has increased tremendously and it poses, according to a closed claim analysis, major risks to patients. Both closed claim analysis identified respiratory depression due to over sedation as the main risk to patients undergoing procedures under sedation. The major problem is that hypoventilation is only detected at very late stages in patients receiving supplemental oxygen. Besides the respiratory effects of hypoventilation, hypercapnia can also lead to hypertension, tachycardia, cardiac arrhythmias and seizures.

The incidence of anesthetized patients with obstructive sleep apnea has increased substantially over the last years along with the current national obesity epidemic. These patients are at increased risk of hypoventilation when exposed to anesthetic drugs. The context of the massive increase in procedural sedation and the extremely high prevalence of obstructive sleep apnea poses major respiratory risks to patients and it may, in a near future, increase malpractice claims to anesthesiologists. The development of safer anesthesia regimen for sedation are, therefore, needed. The establishment of safer anesthetics regimen for sedation is in direct relationship with the anesthesia patient safety foundation priorities. It addresses peri-anesthetic safety problems for healthy patient's. It can also be broadly applicable and easily implemented into daily clinical care. Ketamine has an established effect on analgesia but the effects of ketamine on ventilation have not been clearly defined. The investigators have demonstrated that the transcutaneous carbon dioxide monitor is accurate in detecting hypoventilation in patients undergoing deep sedation. Animal data suggest that when added to propofol in a sedation regimen, ketamine decreased hypoventilation when compared to propofol alone. It is unknown if ketamine added to a commonly used sedative agent (propofol) and fentanyl can decrease the incidence and severity of hypoventilation in patients undergoing deep sedation.

The investigators hypothesize that patients receiving ketamine, propofol and fentanyl will develop less intraoperative hypoventilation than patients receiving propofol and fentanyl.

The investigators also hypothesize that this effect will be even greater in patients with obstructive sleep apnea than patients without obstructive sleep apnea.

Significance: Respiratory depression due to over sedation was identified twice as the major factor responsible for claims related to anesthesia. The high prevalence of obstructive sleep apnea combined with more complex procedures done in outpatient settings can increase physical risks to patients and liability cases to anesthesiologists. The main goal of this project is to establish the effect of ketamine in preventing respiratory depression to patients undergoing procedures under deep sedation using propofol and fentanyl.

If the investigators can confirm our hypothesis, our findings can be valuable not only to anesthesiologist but also to other specialties (emergency medicine, gastroenterologists, cardiologists, radiologists) that frequently performed procedural sedation.

The research questions is; does the addition of ketamine prevent hypoventilation during deep sedation using propofol and fentanyl?

The hypotheses of this study: Ketamine will prevent hypoventilation during deep sedation cases.

ELIGIBILITY:
Inclusion Criteria:

ASA I and II

* Age 18-64
* Females undergoing sedation procedures

Exclusion Criteria:

* Pregnant subjects
* Breastfeeding
* Patients or surgeon request
* Difficult airway

Drop Out:

* Patient or surgeon request
* Conversion to general anesthesia .Inability to obtain data from CO2 monitor.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The total percentage time patients hypoventilate during the case | Day 1
  The total percentage time patients hypoventilate during the case

CONTACTS AND LOCATIONS:
Overall Officials: Gildasio De Oliveira, MD,MS, Principal Investigator — Northwestern University
Locations (1):
- Prentice Womens Hospital, Chicago, Illinois, United States